CLINICAL TRIAL: NCT02564146
Title: Induction Treatment With Nab-paclitaxel/Gemcitabine for First-line Treatment of Metastatic Pancreatic Cancer Followed by Either Alternating Application of Gemcitabine Monotherapy and Nab-paclitaxel/Gemcitabine or Continuing Application of Nab-paclitaxel/Gemcitabine: A Randomized Phase II Study
Brief Title: First-line Treatment of Metastatic Pancreatic Cancer With Nab-paclitaxel and Gemcitabine
Acronym: ALPACA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: ClinAssess GmbH (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIO-PAK-0114; 2014-004086-24 (EudraCT Number); AX-CL-PANC-AIO-004415 (Other Grant/Funding Number: Celgene)
Record Dates: First submitted 2015-09-29; First posted 2015-09-30 (Estimated); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Metastatic Pancreatic Cancer; Adenocarcinoma of the Pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nab-paclitaxel and gemcitabine (A) (Active Comparator): Induction treatment: 3 cycles nab-paclitaxel and gemcitabine
  Continuous treatment after randomization: Continuing application of nab-paclitaxel and gemcitabine treatment cycles
  Interventions: Drug: nab-paclitaxel and gemcitabine
- gemcitabine monotherapy and nab-paclitaxel and gemcitabine (B) (Experimental): Induction treatment: 3 cycles nab-paclitaxel and gemcitabine
  Continuous treatment after randomization: alternating application of gemcitabine monotherapy and nab-paclitaxel and gemcitabine treatment cycles
  Interventions: Drug: nab-paclitaxel and gemcitabine; Drug: gemcitabine mono and nab-paclitaxel and gemcitabine

INTERVENTIONS:
Drug: nab-paclitaxel and gemcitabine — Induction treatment:
  3 cycles nab-paclitaxel and gemcitabine 125 mg/m^2, IV infusion over 30 minutes, followed by gemcitabine 1000 mg/m^2 as a 30-minute IV infusion; D1, D8, D15 of each 28-day cycle.
  Continouous treatment after randomization:
  Continuing application of nab-paclitaxel and gemcitabine treatment cycles until progression or unacceptable toxicity. Duration of each cycle is 28 days nab-paclitaxel 125 mg/m^2, IV infusion over 30 minutes, followed by gemcitabine 1000 mg/m^2 as a 30-minute IV infusion; D1, D8, D15 of each 28-day cycle.
Drug: gemcitabine mono and nab-paclitaxel and gemcitabine — Induction treatment:
  3 cycles nab-paclitaxel and gemcitabine 125 mg/m^2, IV infusion over 30 minutes, followed by gemcitabine 1000 mg/m^2 as a 30-minute IV infusion; D1, D8, D15 of each 28-day cycle.
  Continouous treatment after randomization:
  Alternating application of gemcitabine monotherapy and nab-paclitaxel and gemcitabine treatment cycles until progression or unacceptable toxicity, starting with a treatment cycle of gemcitabine monotherapy.
  Duration of each cycle irrespective of treatment cycle with gemcitabine monotherapy or treatment with nab-paclitaxel/gemcitabine is 28 days.
  Gemcitabine monotherapy treatment cycle: Gemcitabine 1000 mg/m^2 as a 30-minute IV infusion; D1, D8, D15 of each 28-day cycle.
  Nab-paclitaxel and gemcitabine treatment cycle: Nab-paclitaxel 125 mg/m^2, IV infusion over 30 minutes, followed by gemcitabine 1000 mg/m^2 as a 30-minute IV infusion; D1, D8, D15 of each 28-day cycle.
  Arms: gemcitabine monotherapy and nab-paclitaxel and gemcitabine (B)

SUMMARY:
ALPACA is an interventional, multicentre, open-label, randomized active-controlled phase II trial with two arms.

To estimate the treatment effect on overall survival, feasibility, efficacy and safety of alternating treatment cycles of gemcitabine monotherapy followed by nab-paclitaxel/gemcitabine relative to standard continuing nab-paclitaxel/gemcitabine cycles in first-line treatment for metastatic pancreatic cancer in patients having received 3 cycles of induction therapy with standard nab-paclitaxel/gemcitabine.

DETAILED DESCRIPTION:
ALPACA is an interventional, multicentre, open-label, randomized active-controlled phase II trial with two arms.

To estimate the treatment effect on overall survival, feasibility, efficacy and safety of alternating treatment cycles of gemcitabine monotherapy followed by nab-paclitaxel/gemcitabine relative to standard continuing nab-paclitaxel/gemcitabine cycles in first-line treatment for metastatic pancreatic cancer in patients having received 3 cycles of induction therapy with standard nab-paclitaxel/gemcitabine.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years of age)
* Histologically or cytologically confirmed metastatic adenocarcinoma of the pancreas. Patients with islet cell neoplasms are excluded.
* Karnofsky Perfomance Status (KPS) ≥ 70%
* At least one unidimensionally measurable lesion as assessed by CT- scan or Magnetic resonance imaging (MRI) according to Response Evaluation Criteria In Solid Tumors (RECIST1.1 ),
* Total bilirubin ≤ 1.5 x ULN (Upper Limit of Normal). Patients with a biliary stent may be included provided that bilirubin level after stent insertion decreased to ≤ 1.5 x ULN and there is no cholangitis.
* Adequate renal, hepatic and bone marrow function, defined as

  * Calculated creatinine clearance ≥ 30 mL/min according to CKD-EPI formula (Chronic kidney Disease Epidemiology Collaboration)
  * AST/GOT and/or ALT/GPT ≤ 2.5 x ULN and ≤ 5.0 x ULN in case of liver metastasis
  * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
  * Haemoglobin ≥ 9 g/dL
  * Platelets ≥ 100 x 100 x 10^9/L
* Females of Childbearing Potential (FCBP) must have a negative serum pregnancy test within 7 days of the first application of study treatment and they must agree to undergo further pregnancy tests before randomization and at the end of treatment visit and
* FCBP must either agree to use and be able to take effective contraceptive birth control measures (Pearl Index < 1) or agree to practice complete abstinence from heterosexual intercourse during the course of the study and for at least 1 month after last application of study treatment. A female subject is considered to be of childbearing potential unless she is age ≥ 50 years and naturally amenorrhoeic for ≥ 2 years, or unless she is surgically sterile.
* Males must agree not to father a child during the course of the trial and for at least 6 months after last administration of study drugs.
* Signed and dated informed consent before the start of any specific protocol procedures Patient's legal capacity to consent to study participation

Exclusion Criteria:

* Missing histological or cytological confirmation of metastatic adenocarcinoma of the pancreas Locally advanced pancreatic adenocarcinoma without metastases Any previous radiotherapy, surgery, chemotherapy or investigational therapy for the treatment of metastatic disease. (Prior adjuvant chemotherapy with gemcitabine or fluoropyrimidine in curative intent is allowed if terminated more than 6 months before first application of study treatment. Previous palliative radiotherapy of bonemetastases for alleviation of pain is permitted provided that irradiated bone metastases are no target lesions.) Known brain metastase/brain metastases. Brain imaging is required in symptomatic patients to rule out brain metastases, but is not required in asymptomatic patients.
* Pre-existing peripheral neuropathy ≥ grade 2 according to CTCAE version 4 (Common Terminology Criteria for Adverse Events)
* • Medical history of interstitial lung disease (ILD) or pulmonary fibrosis
* Patients with high cardiovascular risk, including, but not limited to, recent coronary stenting or myocardial infarction in the past year.
* Uncontrolled severe illness or medical condition (including uncontrolled diabetes mellitus)
* Any other severe concomitant disease or disorder, which could influence patient's ability to participate in the study and his/her safety during the study or interfere with interpretation of study results e.g. severe hepatic, renal, pulmonary, metabolic, or psychiatric disorders Previous or concurrent tumor other than underlying tumor disease (pancreatic cancer) with the exception of cervical cancer in situ, adequately treated basal cell carcinoma or squamous cell carcinoma of the skin, superficial bladder tumors (Ta, Tis, and T1) or any curatively treated tumors > 5 years prior to enrolment Hypersensitivity against nab-paclitaxel, gemcitabine, or any excipients of these drugs
* Continuing abuse of alcohol, drugs, or medical drugs
* Pregnant females, breast feeding females or females of childbearing potential unable to perform adequate contraceptive measures or practice complete abstinence from heterosexual intercourse
* Participation in any other clinical trial or treatment with any experimental drug within 28 days before enrolment to the study or during study participation until the end of treatment visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2016-12; Primary Completion 2022-03 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | After randomization until date of death or end of study wichever comes first. Assessed for up to 38.5 month
  To estimate the treatment effect of alternating treatment cycles of gemcitabine monotherapy followed by nab-paclitaxel/gemcitabine relative to standard continuing nab-paclitaxel/gemcitabine treatment cycles in first-line treatment for metastatic pancreatic cancer in patients having received 3 cycles of induction therapy with standard nab-paclitaxel/gemcitabine.

SECONDARY OUTCOMES:
Overall survival (OS) | 3.5 month
  During induction phase.
Overall survival (OS) | 42 month
  Determined from first application of induction treatment.
Progression-free survival (PFS) | 3.5 month
  During induction phase.
Progression-free survival (PFS) | Assessed for up to 38.5 month
  As time from randomization to objective tumor progression or death from any cause.
Progression-free survival (PFS) | Assessed for up to 42 month
  As time from randomization to objective tumor progression or death from any cause.
Overall response rate (ORR) | Assessed for up to 42 month
  According to RECISTv1.1 determined from first application of induction treatment.
Overall response rate (ORR) | Assessed for up to 3.5 month
  During induction phase.
Disease control rate (DCR) | Assessed for up to 42 month
  According to RECISTv1.1 determined from first application of induction treatment.
Disease control rate (DCR) | Assessed for up to 3.5 month
  During induction phase.
Quality of life QLQ-C30 | Assessed for up to 3.5 month
  During induction phase.
Quality of life QLQ-C30 | Assessed for up to 8 month
  As determined with EORTC QLQ-C30 determined from randomization.
Adverse Events (AE) | Assessed for up to 11.5 month
  Type, incidence, and severity according to NCI CTCAE version 4 with explicit consideration of any neurotoxicity.
Adverse Events (AE) | Assessed for up to 3.5 month
  Type, incidence, and severity according to NCI CTCAE version 4 with explicit consideration of any neurotoxicity during induction phase.
Time of treatment without toxicity | Assessed for up to 11.5 month
  Duration of treatment without toxicity leading to permanent discontinuation during induction and randomized phase.
Time of treatment without toxicity | Assessed for up to 3.5 month
  Duration of treatment during induction phase.
Neurotoxicity Assessment FACT taxane score | Assessed for up to 11.5 month
  Functional assessment of neurotoxicity (with FACT taxane score) during induction and randomized phase.
Neurotoxicity Assessment FACT taxane score | Assessed for up to 3.5 month
  Functional assessment of neurotoxicity (with FACT taxane score) during induction phase.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Kullmann, Prof. Dr., Principal Investigator — Kliniken Nordoberpfalz AG Klinikum Weiden Medizinische Kliniken I
Locations (1):
- Kliniken Nordoberpfalz AG, Klinikum Weiden, Weiden, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dorman K, Boeck S, Caca K, Reichert M, Ettrich TJ, Oettle H, Waidmann O, Modest DP, Muller L, Michl P, Kanzler S, Pink D, Reinacher-Schick A, Geissler M, Pelz H, Kunzmann V, Held S, Schichtl T, Heinemann V, Kullmann F. Alternating gemcitabine plus nab-paclitaxel and gemcitabine alone versus continuous gemcitabine plus nab-paclitaxel after induction treatment of metastatic pancreatic cancer (ALPACA): a multicentre, randomised, open-label, phase 2 trial. Lancet Gastroenterol Hepatol. 2024 Oct;9(10):935-943. doi: 10.1016/S2468-1253(24)00197-3. Epub 2024 Aug 16. PMID 39159648